CLINICAL TRIAL: NCT07107854
Title: EVALUATION OF THE EFFICACY OF COSMETIC PRODUCT IN ADULTS SUBJECTS WITH MILD TO MODERATE ACNE - USE TEST UNDER DERMATOLOGICAL CONTROL - MULTICENTER STUDY
Brief Title: EVALUATION OF THE EFFICACY OF COSMETIC PRODUCT IN ADULTS SUBJECTS WITH MILD TO MODERATE ACNE
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Other Study IDs: 22E3856 / LRP 22027
Record Dates: First submitted 2025-07-10; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: cosmetic: EFFACLAR ULTRA CONCENTRATED SERUM — Transparent solution (gel)

SUMMARY:
EVALUATION OF THE EFFICACY OF COSMETIC PRODUCT IN ADULTS SUBJECTS WITH MILD TO MODERATE ACNE. USE TEST UNDER DERMATOLOGICAL CONTROL. THE STUDY CONDUCTED IN POLAND AND MAURITIUS

DETAILED DESCRIPTION:
Claims:

* Improvement of acne
* Improvement of skin smoothness parameters

Objectives:

To evaluate:

* Its capacity to maintain the human face in good condition (cutaneous acceptability) by clinical examination under dermatological control;
* their comedogenic potential by counting the retentional and inflammatory lesions by the dermatologist in charge of the study;
* its smoothing effect by collecting polymer silicone skin's prints Silflo® and analysis using 3D Primos® Compact System
* its capacity to improve skin elasticity using cutometer®
* its capacity to maintain skin hydration using corneometer®
* its effect on the skin state by clinical scoring by the dermatologist in charge of the study;
* its effect on skin state by clinical auto scoring by the subjects;
* their anti-acne effect by GEA score and AFAST (score B) by the dermatologist in charge of the study;
* to illustrate their visual expected effect using ColorFace® and skincam®;
* to evaluate the change of subjects' quality of life questionnaire (AI-ADL) from baseline to D84 and D168;
* subjectively its cosmetic acceptability, properties, efficacy and future use by analysis of the subjects' answers to a subjective evaluation questionnaire

ELIGIBILITY:
Inclusion Criteria:

- Sex: female and male;

* Age: 20 years old and above;
* Type: Caucasian;
* Phototype: I to VI
* At least 10 subjects per phototype;
* At least 5 subjects with GEA 3 per phototype;
* At least 2 males per phototype
* Subjects with mild to moderate acne (GEA 2-3);
* Subjects with at least 8 inflammatory lesions (full face);
* Subjects at least 20 non inflammatory lesions (full face). Healthy subject;
* Subject having given her/his free informed, web written consent;
* Subject willing to adhere to the protocol and study procedures.

Exclusion Criteria:

* Concerns woman: Pregnant or nursing woman or woman planning to get pregnant during the study;

  * Cutaneous pathology on the studied zone other than acne (eczema etc.);
  * Use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the acceptability and efficacy of the studied products (according to the investigator's appreciation);
  * Oral treatment of retinoids during the six previous months of the study;
  * Topical acne treatment since less than one month;
  * Acne with documented hormonal origin (e.g PCOS, hyperandrogenia of other origin).
  * Any change in hormonal treatment (including contraceptive) during the three previous months of the study or subject under Androcur®;
  * Subject under cyproterone-based or drospirenone medications (like Diane 35®, or Jasmine®, or Holgyème® or generic) treatments since less than six months;
  * Professional facial care during the previous month of the study;
  * Subject manipulating her acne lesions;
  * Subject with make-up on the day of the visit at the laboratory;
  * Excessive exposure to sunlight or UV-rays within the previous month;
  * Subject having undergone a surgery under general anesthesia within the previous month;
  * Subject enrolled in another clinical trial during the study period (concerns the studied zone);
  * Subject considered by the investigator to be likely not compliant to the protocol;
  * Subject enrolled in another clinical trial during the study period (concerns the studied zone);
  * Subject who does not meet the Ministry of Health guidelines for COVID-19 at time of the visit.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sex: female and male;
  * Age: 20 years old and above;
  * Type: Caucasian;
  * Phototype: I to VI
  * At least 10 subjects per phototype;
  * At least 5 subjects with GEA 3 per phototype;
  * At least 2 males per phototype
  * Subjects with mild to moderate acne (GEA 2-3);
  * Subjects with at least 8 inflammatory lesions (full face);
  * Subjects at least 20 non inflammatory lesions (full face). Healthy subject;
  * Subject having given her/his free informed, web written consent;
  * Subject willing to adhere to the protocol and study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
comedogenic potential | kinetics: Day 0, Day 14, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
  comedogenic potential by counting the retentional and inflammatory lesions by the dermatologist in charge of the study;

CONTACTS AND LOCATIONS:
Locations (1):
- PAŁUBICKA Joanna, Gdansk, Gdańsk, Poland

IPD SHARING:
Plan to Share IPD: No